CLINICAL TRIAL: NCT00034177
Title: Safety And Efficacy Of Weekly Administration Of S-8184 Paclitaxel Injectable Emulsion In Second Line Treatment Of Patients With Locally Advanced, Metastatic, Or Recurrent Transitional Cell Carcinoma Of The Urothelium
Brief Title: Safety and Efficacy of S-8184 in Treatment of Locally Advanced, Metastatic, or Recurrent TCC of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Monica Krieger, VP Regulatory Affairs, OncoGenex Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SON-8184-1065
Record Dates: First submitted 2002-04-23; First posted 2002-04-25 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Urologic Neoplasms
Keywords: Locally Advanced, Metastatic, or Recurrent Transitional Cell Carcinoma of the Urothelium
MeSH Terms: conditions — Urologic Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: S-8184 Paclitaxel Injectable Emulsion
Drug: Experimental Arm: TOCOSOL Paclitaxel — Doses of 80, 100 and 120mg/m2

SUMMARY:
Phase IIA, multicenter, dose escalation study evaluating the safety and efficacy of weekly S-8184 paclitaxel injectable emulsion in second line treatment of patients locally advanced, metastatic, or recurrent transitional cell carcinoma of the urothelium.

DETAILED DESCRIPTION:
The goals of this study are to determine the objective response rate, to determine time to disease progression, duration of response, and survival, and to identify the maximum tolerated weekly dose and principal toxicities of S-8184 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of transitional cell carcinoma of the urothelium including renal pelvis, ureter, bladder, or urethra
* Locally advanced with lymph node disease(unresectable T3-4, N+, M0); metastatic (T any, N any, MI); or locally recurrent disease following initial definitive therapy
* One and only one prior systemic cytotoxic chemotherapy regimen (note that intravesical treatments are not included in the definition of systemic cytotoxic chemotherapy)
* Failure of first line systemic chemotherapy with a platinum-containing combination regimen consisting of MVAC or cisplatin/gemcitabine with cisplatin dosed at 60 mg/m2 or higher per cycle
* Adult (18 years of age or older) patients
* Adequate hematologic function (ANC greater than 1500 cells/mm3 and platelets greater than 100,000/mm3)
* Serum creatinine less than 2.0 mg/dL
* Total bilirubin less than 1.5 mg/dL; SGOT and SGPT less than 3 times the upper limit of institutional normal values
* ECOG performance status of 0 - 2
* Bidimensional measurable disease
* Patients who have signed an IRB / Ethics Committee approved informed consent
* Life expectancy at least 12 weeks
* Patient has fully recovered from any previous surgery (at least 4 weeks since major surgery)
* Patient has a negative pregnancy test prior to study entry if premenopausal. (Patients of child bearing potential must use a medically effective form of contraception during the treatment.)

Exclusion Criteria:

* Patients who have received any taxane-containing preparation including Taxol (paclitaxel) or Taxotere (docetaxel)
* Patients with intracranial metastases
* Females who are pregnant or lactating
* Patients with peripheral neuropathy NCI-CTC grade 2 or greater
* Patients who have received wide-field radiation, cytotoxic chemotherapy or hormonal therapy within 4 weeks of study entry; or mitomycin or nitrosoureas within 6 weeks of study entry
* Patients who have had an investigational agent within 4 weeks of study entry
* Patients receiving concurrent anticonvulsants known to induce P450 isoenzymes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate; time to disease progression; duration of response; survival; toxicities | After all patients completed treatment

SECONDARY OUTCOMES:
To determine time to disease progression | After all patients have completed treatment